CLINICAL TRIAL: NCT01649427
Title: Multi-center, Open-label, Prospective, Randomized, Parallel Group Study Investigating a Tacrolimus Hexal® Based Regimen Versus a Prograf® Based Regimen in de Novo Renal Transplant Recipients
Brief Title: Comparison of a Tacrolimus Hexal® Based Regimen Versus a Prograf® Based Regimen in de Novo Renal Transplant Recipients
Acronym: Spartacus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CERL080ADE27
Record Dates: First submitted 2012-07-20; First posted 2012-07-25 (Estimated); Results first posted 2019-06-17 (Actual); Last update posted 2019-06-17 (Actual); Status verified 2017-11

CONDITIONS: Pharmacokinetics Study in de Novo Kidney Transplantation
Keywords: Pharmacokinetics Study; Tacroliums; GFR; kidney; transplant rejection; allograft rejection; xenograft rejection; host vs graft disease; renal transplant
MeSH Terms: conditions — Graft vs Host Disease | interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prograf (Experimental): Control therapy: one capsule containing 0.5 mg, 1mg or 5mg Prograf®, one tablet containing 180mg or 360mg Myfortic®, corticosteroids and one vial containing 20mg lyophilisate Simulect®
  Interventions: Drug: Prograf
- Tacroliums Hexal (Experimental): Investigational therapy: one capsule containing 0.5mg, 1mg or 5mg Tacrolimus Hexal®, one tablet containing 180mg or 360mg Myfortic®, corticosteroids and one vial containing 20mg lyophilisate Simulect®
  Interventions: Drug: Tacrolimus Hexal

INTERVENTIONS:
Drug: Prograf — Prograf® capsules were supplied as capsules of 0.5 mg, 1 mg and 1.5 mg dose strengths.
  Arms: Prograf
Drug: Tacrolimus Hexal — Tacrolimus Hexal® capsules were supplied to the investigators at dose strengths of 0.5 mg,
  1 mg and 1.5 mg.
  Arms: Tacroliums Hexal

SUMMARY:
The purpose of this study was to investigate if Tacrolimus Hexal® has similar pharmacokinetic properties compared to Prograf® in de novo renal transplant patients and whether the comparable exposure resulted in similar renal function.

DETAILED DESCRIPTION:
In Phase II of this study there was a high patient drop-out rate and an associated long recruitment timespan. Eighty-one patients were recruited to Phase I and only 45 of the required 54 patients were available for PK analysis. To complete Phase II, 245 (in addition to 81) patients were to be required to achieve calculated sample size. Therefore the protocol was amended to stop recruitment and analyze Phase I patient data of CERL080ADE27 (PK-Phase I). Patients that were still ongoing were scheduled for an end of study (EOS) visit. During this visit patients were informed by the investigator about the end of study and advised about further treatment course.

ELIGIBILITY:
Inclusion:

primary or sec. kidney transplanted patiens, written consent, cold ischemia < 24 h

Exclusion:

multi organ, immunological risc pts., PRA >20%, Antibodys against HLA-type of donor organ, hypersensitivity against Tacro or MMF,

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 73 (Actual)
Dates: Start 2012-10-17 (Actual); Primary Completion 2015-08-20 (Actual); Study Completion 2015-08-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (5):
- Germany (5):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bochum
  - Novartis Investigative Site, Düsseldorf
  - Novartis Investigative Site, Kaiserslautern
  - Novartis Investigative Site, Koeln-Merheim

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 81 patients were randomized, but only 73 were assigned drug. 1 patient who was excluded from efficacy analyses, was randomized to Prograf but did not receive treatment but kept for safety reporting. 74 patients were used for safety analysis while only 73 were available for efficacy analysis
Pre-assignment Details: This is a 2-phase study:
  PHASE I:
  In 1st phase of study, PK parameters were evaluated in total of 60 evaluable patients (30 patients per treatment group)
  Phase II was not conducted
Groups:
- Tacrolimus Hexal®: Investigational therapy: one capsule containing 0.5mg, 1mg or 5mg Tacrolimus Hexal®, one tablet containing 180mg or 360mg Myfortic®, corticosteroids and one vial containing 20mg lyophilisate Simulect®
- Prograf®: Control therapy: one capsule containing 0.5 mg, 1mg or 5mg Prograf®, one tablet containing 180mg or 360mg Myfortic®, corticosteroids and one vial containing 20mg lyophilisate Simulect®
Period: Overall Study
Arm/Group | Tacrolimus Hexal® | Prograf®
Started | 35 | 38
Completed | 24 | 26
Not Completed | 11 | 12
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 8 | 7
Not completed — Lost to Follow-up | 0 | 1
Not completed — Graft loss | 0 | 1
Not completed — Surgical problems during nephrectomy | 2 | 2

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) consisted of all patients in whom study treatment was assigned. Following the intent-to-treat principle, patients were analyzed according to the treatment they were assigned to at randomization
Groups:
- Total: Total of all reporting groups
Arm/Group | Tacrolimus Hexal® | Prograf® | Total
Number analyzed (Participants) | 35 | 38 | 73
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.9 (9.9) | 47.2 (11.8) | 47.5 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 9 | 15
  Male | 29 | 29 | 58

OUTCOME MEASURES:

1. Primary Outcome: ANCOVA Model for Change in Nankivell GFR (mL/Min) at Month 6, Without Replacement of Missing Values (Full Analysis Set)
Description: Change in Nankivell glomerular filtration rate (GFR) from baseline to 6 months
  Glomerular Filtration Rate (GFR): The GFR is the best clinical estimate of renal function in health and disease, and correlates well with the clinical severity of renal function disturbances. Several studies have shown that in patients with progressive renal disease, GFR declines or reciprocal serum creatinine levels elevate linearly over time in a predictable manner. With the help of the serum creatinine values, the GFR was calculated via Nankivell formula.
Time Frame: baseline to month 6
Population: as for baseline characteristics
Measure: Least Squares Mean (95% Confidence Interval); unit: mL/min
Arm/Group | Tacrolimus Hexal® | Prograf®
Number analyzed (Participants) | 24 | 27
mL/min | 47.65 (20.24) [41.70 to 53.60] | 38.60 (18.83) [31.32 to 45.89]
Statistical Analysis 1: Comparison: Tacrolimus Hexal® vs Prograf®; Test type: Non-Inferiority or Equivalence — Non-inferiority; p = 0.0003, ANCOVA

2. Secondary Outcome: The Incidence of Biopsy-proven Acute Rejection (BPAR), Graft Loss and Death Until Month 12 (Full Analysis Set) (Full Analysis Set)
Description: The key secondary objective was to assess the incidence of individual endpoints BPAR, graft loss and death until month 6 post-transplantation.
Time Frame: baseline to month 12
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Incidences
Arm/Group | Tacrolimus Hexal® | Prograf®
Number analyzed (Participants) | 35 | 38
Incidences
  Biopsy proven acute rejection (BPAR) | 2 [0.70 to 19.16] | 3 [1.66 to 21.38]
  Graft loss | 0 [0.00 to 10.00] | 1 [0.07 to 13.81]
  Death | 0 [0.00 to 10.00] | 1 [0.07 to 13.81]
  Composite: BPAR, graft loss or death | 2 [0.70 to 19.16] | 4 [2.94 to 24.80]

3. Secondary Outcome: ANCOVA Model for Change in CKD-EPI GFR (Chronic Kidney Disease Epidemiology Collaboration Glomerular Filtration Rate) at Month 6 Post-transplantation
Description: ANCOVA model for change in CKD-EPI Glomerular Filtration Rate (GFR)[ml/min] without replacement of missing values
Time Frame: baseline to Month 6
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: mL/min
Arm/Group | Tacrolimus Hexal® | Prograf®
Number analyzed (Participants) | 24 | 27
mL/min | 48.33 (3.84) | 39.77 (4.61)

4. Primary Outcome: ANOVA for Dose-normalized Tacrolimus 12-h-AUC (h/103*L) at Month 1
Description: Compares the PK of Tacrolimus Hexal® assessed by the ratio of the AUC0-12h over one month period post transplantation vs. Prograf® in renal transplant patients
Time Frame: end of month 1
Measure: Least Squares Mean (90% Confidence Interval); unit: h/10^3*L
Arm/Group | Tacrolimus Hexal® | Prograf®
Number analyzed (Participants) | 23 | 20
h/10^3*L
  Adjusted, log-transformed Estimates (ANOVA) | 2.944 [2.783 to 3.105] | 3.020 [2.811 to 3.228]
  Adjusted, back-transformed Estimates (ANOVA) | 18.991 [16.163 to 22.314] | 20.484 [16.630 to 25.231]

5. Secondary Outcome: ANCOVA Model for Change in MDRD GFR (ml/Min) at Month 6, Without Replacement of Missing Values
Description: MDRD GFR
Time Frame: least square (LS) mean change from baseline to Month 6
Measure: Least Squares Mean (95% Confidence Interval); unit: (ml/min)
Arm/Group | Tacrolimus Hexal® | Prograf®
Number analyzed (Participants) | 35 | 38
(ml/min) | 46.20 [37.62 to 54.79] | 38.52 [28.64 to 48.41]

6. Secondary Outcome: ANCOVA Model for Change in Cockcroft-Gault GFR (ml/Min) at Month 6, Without Replacement of Missing Values
Description: change in Cockcroft-Gault GFR
Time Frame: least square (LS) mean change from baseline to Month 6
Measure: Least Squares Mean (95% Confidence Interval); unit: (ml/min)
Arm/Group | Tacrolimus Hexal® | Prograf®
Number analyzed (Participants) | 35 | 38
(ml/min) | 60.45 [52.48 to 68.41] | 46.45 [36.89 to 56.02]

ADVERSE EVENTS:
Description: One patient was randomized to Prograf but didn't receive assigned treatment hence was excluded from efficacy analyses but was kept for safety reporting
Groups:
- Tacrolimus Hexal: Investigational therapy: one capsule containing 0.5mg, 1mg or 5mg Tacrolimus Hexal®, one tablet containing 180mg or 360mg Myfortic®, corticosteroids and one vial containing 20mg lyophilisate Simulect®
Arm/Group | Tacrolimus Hexal | Prograf
Serious Adverse Events (participants affected / at risk) | 19/35 | 17/39
Other Adverse Events (participants affected / at risk) | 34/35 | 38/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tacrolimus Hexal (N=35) | Prograf (N=39)
LEUKOPENIA (Blood and lymphatic system disorders) | 1 | 1
THROMBOTIC MICROANGIOPATHY (Blood and lymphatic system disorders) | 0 | 2
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 1 | 0
CORONARY ARTERY DISEASE (Cardiac disorders) | 0 | 1
COLITIS (Gastrointestinal disorders) | 1 | 0
DIARRHOEA (Gastrointestinal disorders) | 3 | 0
ENTERITIS (Gastrointestinal disorders) | 0 | 1
LARGE INTESTINE PERFORATION (Gastrointestinal disorders) | 1 | 0
PANCREATIC PSEUDOCYST (Gastrointestinal disorders) | 1 | 0
PANCREATITIS CHRONIC (Gastrointestinal disorders) | 1 | 0
IMPAIRED HEALING (General disorders) | 1 | 0
IMPLANT SITE EXTRAVASATION (General disorders) | 1 | 0
OEDEMA PERIPHERAL (General disorders) | 1 | 0
PYREXIA (General disorders) | 0 | 1
KIDNEY TRANSPLANT REJECTION (Immune system disorders) | 2 | 2
BACTERIAL SEPSIS (Infections and infestations) | 0 | 1
BRONCHITIS (Infections and infestations) | 0 | 1
CAMPYLOBACTER GASTROENTERITIS (Infections and infestations) | 1 | 0
CYTOMEGALOVIRUS INFECTION (Infections and infestations) | 0 | 1
DIVERTICULITIS (Infections and infestations) | 1 | 0
ENTEROCOCCAL INFECTION (Infections and infestations) | 0 | 1
HUMAN POLYOMAVIRUS INFECTION (Infections and infestations) | 0 | 1
INFECTION (Infections and infestations) | 0 | 1
LUNG INFECTION (Infections and infestations) | 1 | 1
PERITONITIS (Infections and infestations) | 1 | 0
POLYOMAVIRUS-ASSOCIATED NEPHROPATHY (Infections and infestations) | 1 | 0
SINUSITIS (Infections and infestations) | 0 | 1
URINARY TRACT INFECTION (Infections and infestations) | 4 | 4
UROSEPSIS (Infections and infestations) | 2 | 0
ABDOMINAL WOUND DEHISCENCE (Injury, poisoning and procedural complications) | 1 | 1
COMPLICATIONS OF TRANSPLANTED KIDNEY (Injury, poisoning and procedural complications) | 4 | 3
DELAYED GRAFT FUNCTION (Injury, poisoning and procedural complications) | 1 | 0
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
INCISIONAL HERNIA (Injury, poisoning and procedural complications) | 2 | 0
TOXICITY TO VARIOUS AGENTS (Injury, poisoning and procedural complications) | 1 | 0
TRAUMATIC HAEMOTHORAX (Injury, poisoning and procedural complications) | 1 | 0
BLOOD CREATININE INCREASED (Investigations) | 4 | 1
DEHYDRATION (Metabolism and nutrition disorders) | 1 | 0
HYPERKALAEMIA (Metabolism and nutrition disorders) | 0 | 1
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 0 | 1
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 3 | 0
DYSURIA (Renal and urinary disorders) | 1 | 0
FOCAL SEGMENTAL GLOMERULOSCLEROSIS (Renal and urinary disorders) | 2 | 0
PROTEINURIA (Renal and urinary disorders) | 3 | 0
RENAL FAILURE (Renal and urinary disorders) | 0 | 1
RENAL IMPAIRMENT (Renal and urinary disorders) | 2 | 1
URETERAL NECROSIS (Renal and urinary disorders) | 0 | 1
URETERIC STENOSIS (Renal and urinary disorders) | 1 | 1
URINARY INCONTINENCE (Renal and urinary disorders) | 0 | 1
URINARY RETENTION (Renal and urinary disorders) | 1 | 0
URINARY TRACT DISORDER (Renal and urinary disorders) | 1 | 0
URINARY TRACT OBSTRUCTION (Renal and urinary disorders) | 0 | 1
URINOMA (Renal and urinary disorders) | 1 | 0
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 | 0
SLEEP APNOEA SYNDROME (Respiratory, thoracic and mediastinal disorders) | 1 | 0
SKIN ULCER (Skin and subcutaneous tissue disorders) | 1 | 0
VARICOSE VEIN (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tacrolimus Hexal (N=35) | Prograf (N=39)
ANAEMIA (Blood and lymphatic system disorders) | 4 | 7
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 0 | 2
LEUKOPENIA (Blood and lymphatic system disorders) | 3 | 7
NEPHROGENIC ANAEMIA (Blood and lymphatic system disorders) | 5 | 2
SINUS TACHYCARDIA (Cardiac disorders) | 1 | 2
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 2
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 | 2
CONSTIPATION (Gastrointestinal disorders) | 2 | 6
DIARRHOEA (Gastrointestinal disorders) | 5 | 5
FLATULENCE (Gastrointestinal disorders) | 3 | 4
HIATUS HERNIA (Gastrointestinal disorders) | 1 | 3
NAUSEA (Gastrointestinal disorders) | 2 | 5
VOMITING (Gastrointestinal disorders) | 1 | 3
IMPAIRED HEALING (General disorders) | 1 | 2
OEDEMA PERIPHERAL (General disorders) | 3 | 7
PYREXIA (General disorders) | 1 | 3
KIDNEY TRANSPLANT REJECTION (Immune system disorders) | 1 | 4
CYTOMEGALOVIRUS INFECTION (Infections and infestations) | 1 | 4
CYTOMEGALOVIRUS VIRAEMIA (Infections and infestations) | 2 | 0
NASOPHARYNGITIS (Infections and infestations) | 2 | 3
PNEUMONIA (Infections and infestations) | 0 | 2
SEPSIS (Infections and infestations) | 0 | 2
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 | 1
URINARY TRACT INFECTION (Infections and infestations) | 6 | 16
WOUND INFECTION (Infections and infestations) | 0 | 2
COMPLICATIONS OF TRANSPLANTED KIDNEY (Injury, poisoning and procedural complications) | 5 | 11
POST PROCEDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 2 | 3
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 2 | 1
RENAL LYMPHOCELE (Injury, poisoning and procedural complications) | 4 | 3
WOUND COMPLICATION (Injury, poisoning and procedural complications) | 16 | 19
WOUND DEHISCENCE (Injury, poisoning and procedural complications) | 2 | 1
BLOOD CREATININE INCREASED (Investigations) | 2 | 6
C-REACTIVE PROTEIN INCREASED (Investigations) | 0 | 2
HEPATIC ENZYME INCREASED (Investigations) | 0 | 3
ACIDOSIS (Metabolism and nutrition disorders) | 0 | 2
DIABETES MELLITUS (Metabolism and nutrition disorders) | 3 | 2
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 1 | 2
HYPERCHOLESTEROLAEMIA (Metabolism and nutrition disorders) | 2 | 1
HYPERKALAEMIA (Metabolism and nutrition disorders) | 9 | 9
HYPERLIPIDAEMIA (Metabolism and nutrition disorders) | 3 | 1
HYPERPHOSPHATAEMIA (Metabolism and nutrition disorders) | 1 | 2
HYPERURICAEMIA (Metabolism and nutrition disorders) | 3 | 9
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 5 | 4
HYPOKALAEMIA (Metabolism and nutrition disorders) | 5 | 4
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 5 | 7
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 3 | 2
IRON DEFICIENCY (Metabolism and nutrition disorders) | 0 | 2
METABOLIC ACIDOSIS (Metabolism and nutrition disorders) | 2 | 3
VITAMIN D DEFICIENCY (Metabolism and nutrition disorders) | 2 | 6
HEADACHE (Nervous system disorders) | 4 | 1
TREMOR (Nervous system disorders) | 3 | 2
INSOMNIA (Psychiatric disorders) | 4 | 6
RESTLESSNESS (Psychiatric disorders) | 0 | 2
SLEEP DISORDER (Psychiatric disorders) | 3 | 1
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 | 2
BLADDER PAIN (Renal and urinary disorders) | 5 | 3
BLADDER SPASM (Renal and urinary disorders) | 0 | 3
OLIGURIA (Renal and urinary disorders) | 0 | 2
RENAL FAILURE (Renal and urinary disorders) | 0 | 2
RENAL HYPERTENSION (Renal and urinary disorders) | 0 | 4
URINARY RETENTION (Renal and urinary disorders) | 2 | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 2
ACNE (Skin and subcutaneous tissue disorders) | 2 | 0
ALOPECIA (Skin and subcutaneous tissue disorders) | 0 | 2
SCAR PAIN (Skin and subcutaneous tissue disorders) | 0 | 2
HYPERTENSION (Vascular disorders) | 12 | 20

LIMITATIONS AND CAVEATS:
1 patient was randomized to Prograf but didn't get treatment and was excluded from efficacy analyses but kept for safety reporting. Phase 2 was not started due to high drop-out rate. 73 enrolled; 43 of the planned 54 were available for PK analysis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial